CLINICAL TRIAL: NCT00781313
Title: Pre-hurricane Disaster Preparedness: A Survey in Pediatric Type 1 Diabetes
Brief Title: Disaster Preparedness Among Families Caring for Children With Diabetes
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rubina Heptulla, MD, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-23261
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim of the survey is to ascertain the emergency preparedness among our families with diabetes mellitus and to obtain a percentage of unprepared to the ones who are prepared. The secondary aim is to demonstrate the relationship between disaster preparedness and factors like socio-economic status, parent's marital status, ethnicity and those who had prior experience of a disaster to those who have not experienced a disaster.

DETAILED DESCRIPTION:
This is a cross-sectional study. The subjects are the parent/parents/legal guardian, who will be coming to the clinic for their routine appointment for diabetes management. During the time in which the subject is waiting for the doctor or after their check-up, a research team member will approach the family and ask for their permission to administer the survey. The survey consists of a series of questions designed to ascertain the awareness towards emergency preparedness among families. After they have completed the questionnaire they would be given and/or mailed handouts to enhance their awareness towards disaster preparedness.

Potential Benefits:

This study will help to increase awareness regarding disaster preparedness among the surveyed families. Subjects and families will gain valuable information about caring for diabetes in the event of a disaster.

The potential benefit to the society is that through this study we can ascertain the primary caregiver's awareness of disaster preparedness in regard to a family member with a chronic illness. We will suggest measures to improve their competency towards dealing with disasters. We will be providing educational literature to the primary care givers in the form of handouts at the end of the survey.

ELIGIBILITY:
Inclusion Criteria:

* Subjects include families of children with type 1 and type 2 diabetes mellitus attending the Diabetes/ Endocrine Clinic at Texas Children Hospital.

Exclusion Criteria:

* Subjects excluded are families of Children with illnesses other than type 1 and type 2 diabetes mellitus attending the Diabetes/ Endocrine Clinic at Texas Children Hospital.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target populations for our study are the families attending the Diabetes/ Endocrine Clinic at Texas Children Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary aim is to ascertain the emergency preparedness among our families with diabetes mellitus and to obtain a percentage of unprepared to the ones who are prepared. | September 2008

CONTACTS AND LOCATIONS:
Overall Officials: RUBINA A HEPTULLA, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No